CLINICAL TRIAL: NCT07277582
Title: A Phase 2/3, Two-part, Dose-ranging, Adaptive Study to Evaluate Efficacy and Safety of THRV-1268 in Participants Diagnosed With Long QT Syndrome Type 2 (LQTS 2)
Brief Title: Evaluation of Efficacy and Safety of THRV-1268 in Long QT Syndrome Type 2 (LQTS 2)
Acronym: Wave II
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Thryv Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THRV-1268-0392
Record Dates: First submitted 2025-12-02; First posted 2025-12-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Long QT Syndrome (LQTS) 2
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- THRV-1268 (Experimental): 3 weeks lead-in baseline followed by 50 mg BID for 6 weeks with scheduled up-titration to 100 mg BID for another 6 weeks (12 weeks total treatment)
  Interventions: Other: baseline lead-in; Drug: THRV-1268

INTERVENTIONS:
Other: baseline lead-in — Participants will undergo a 3 weeks run-in baseline
Drug: THRV-1268 — THRV-1268 50 mg bid (total daily 100 mg) for 6 weeks
Drug: THRV-1268 — THRV-1268 100 mg bid (total daily 200 mg) for 6 weeks

SUMMARY:
The goal of this clinical trial is to learn whether the study drug THRV-1268 can safely and effectively shorten the QT interval in people diagnosed with Long QT Syndrome Type 2 (LQTS 2). The study will also learn about the safety and tolerability of THRV-1268 at different doses.

The main questions this study aims to answer are:

Does THRV-1268 reduce the QTc interval (a measure of the heart's electrical recovery time)?

What side effects or medical problems occur when participants take THRV-1268?

Which dose of THRV-1268 works best and is safest?

Participants will:

Complete a 3-week observation period with ECG and Holter monitoring to establish baseline QTc measurements Take THRV-1268 tablets twice daily at two dose levels for 6 weeks (Part A) or be randomly assigned to a dose group for 6 weeks (Part B)

Have clinic visits and tests to monitor safety and changes in their heart rhythm

May continue taking THRV-1268 for up to 1 year for ongoing safety and efficacy evaluation

Researchers will compare changes in QTc over time and evaluate side effects to determine whether THRV-1268 can help reduce the risk of abnormal heart rhythms and sudden cardiac events in people with LQTS 2.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants over 15 years of age at Screening (at least the first 5 participants enrolled in Part A must be 18 years of age or older).
* LQTS 2 genotype: Demonstration of KCNH2 mutation by clinical laboratory test result that is autosomal dominant (heterozygous) and considered to be pathologic or likely pathologic can be included after approval from the sponsor medical monitor or qualified delegate.
* QTcF interval >480 ms and ≤600 ms based on Screening ECG.
* Body weight of at least 45 kg with body mass index between 18.0 and 40.0 kg/m2, inclusively at Screening.
* Male and female participants of childbearing potential must agree to use highly effective contraception throughout the duration of the study.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Participants age 15 to <18 years capable of providing signed assent.

Exclusion Criteria:

* Within 2 months prior to Screening, Participant has a history of an aborted cardiac arrest, ICD implantation, or syncopal episode due to a ventricular arrhythmia. Participants can be enrolled after the 2-month period has lapsed.
* History of structural or functional cardiovascular disease, myocardial infarction or stroke or transient ischemic attack (TIA), atrial fibrillation or atrial flutter, heart failure, bundle branch block, angina pectoris, or hemodynamically significant ventricular tachycardia not due to TdP
* Active or known liver disease.
* Active or past oncologic disease, except for non-melanoma skin cancer.
* Advanced pulmonary disease that requires more than a steroid inhaler.
* Pulmonary artery hypertension.
* Is pregnant, lactating, or breastfeeding, or planning to become pregnant.
* Has a positive result for the urine pregnancy test at the Screening Visit or the serum pregnancy test at the Day -7 Visit.
* Clinically significant abnormal findings on the physical examination or medical history during Screening or Day -21 as deemed by the investigator.
* Has experienced an acute illness that has resolved in less than 14 days before the first study drug dose or has had a major illness or hospitalization within 1 month before the first study drug dose.
* Has a recent history of alcohol or substance abuse that would pose a risk for the participant's safety and compliance with the study protocol, in the opinion of the investigator.
* Has a pacemaker or ICD that is actively used for ventricular pacing.
* Is currently taking or anticipates the use of any restricted drugs
* Is considering or scheduled to undergo any elective surgical procedure during the study.
* Current participation or recent within 1 month of participating in another interventional clinical study.
* Screening Visit diastolic blood pressure >95 mm Hg, systolic blood pressure <90 or >150 mm Hg.
* At Screening, if the 12-lead triplicate ECG demonstrates any of the following: PR >280 ms; QRS >110 ms, or QTcF >600 ms or ≤480 ms; bundle branch block or significant ST-T wave abnormalities or flat T waves that could interfere with QT analysis. HR <50 bpm, unless receiving a beta-blocker in which case <40 bpm, or HR >100 bpm at rest.
* Atrial pacing rate set to >80 bpm in those participants with atrial pacing.
* Abnormal renal function with an eGFR of <70 mL/min/1.73 m2 (with eGFR calculated by the CKD-EPI formula at Screening). One retest of the exclusionary eGFR value is allowed at the discretion of the investigator.
* Has abnormal liver function tests:

  * ALT, AST, GGT, ALP > 1.5 the ULN.
  * Total bilirubin >ULN.
  * INR >1.2 ULN (requires measurement of prothrombin time (PT)).
* Has clinically significant abnormality in serum chemistry values at Screening for hemoglobin, potassium, magnesium, or calcium levels as determined by the investigator. A single repeat test and/or correction of abnormal values (e.g., electrolyte repletion) is permitted at the investigator's discretion prior to enrollment.
* Any participant, who, for any reason, is deemed by the investigator to be inappropriate for this study or has any condition which would confound or interfere with the evaluation of the safety, tolerability, or efficacy of the investigational medicinal product (IMP) or prevent compliance with the study protocol.
* Consumes on average more than 21 standard alcoholic drinks per week in men and 14 standard drinks per week in women over the last 2 years.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Part A: To evaluate the effect of oral THRV-1268 on QTcF interval by AUC method in participants with LQTS 2 | Day 42 and Day 84
  ΔAUC0-6 hours QTcF values on Day 42 (THRV-1268 50 mg BID) and Day 84 (THRV-1268 100 mg BID) compared to the the baseline (mean of Day -7 and Day -1).
Part A: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | up to 52 weeks
  To assess the safety and tolerability of two oral dose levels of THRV-1268 in participants with LQTS2 by measuring the incidence of treatment-emergent adverse events throughout the study.

SECONDARY OUTCOMES:
Part A: To evaluate the effects of oral THRV-1268 on QTcF interval by various methods in participants with LQTS 2 | from 0 to 12 hours on Day 42 and 84
  QTcF values at each timepoint on Days 42 and 84 will be compared to the time-matched QTcF values on Baseline (mean of Day -7 and Day -1).
Part A: To evaluate the effect of oral THRV-1268 on QTcF interval by AUC method in participants with LQTS 2 | Day 42 and Day 84
  ΔAUC0-12/12 QTcF values on Day 42 (THRV-1268 50 mg BID) and Day 84 (THRV-1268 100 mg BID) compared to the the baseline (mean of Day -7 and Day -1).
Part A: To evaluate the effect of oral THRV-1268 on QTcF interval by AUC method in participants with LQTS 2 | Day 42 and Day 84
  ΔAUC0-6 hours QTcF values on Day 42 (THRV-1268 50 mg BID) and Day 84 (THRV-1268 100 mg BID) compared to the the baseline (mean of Day -7 and Day -1) in patients with mean baseline AUC(0-6)/6 QTcF >500 ms.
Part A: To evaluate the maximal shortening in QTcF from pre-dose to post-dose | Day 42 and Day 84
  Measure the maximum delta between pre-dose QTcF (mean baseline values at Day-7 and Day-1) and lowest QTcF values reported on Day 42 and Day 84.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Honor Health Research and Innovation Institute, Scottsdale, Arizona
  - University of California San Francisco, San Francisco, California
  - University of Illinois Chicago, Chicago, Illinois
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Heart Center Clinical Research Program | MGH, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Rochester Medical Center, Rochester, New York
  - Wilmington Health, Wilmington, North Carolina